CLINICAL TRIAL: NCT03444792
Title: Mechanical Dilatation vs Non-Dilatation of the Cervix at Elective Caesarean Section to Reduce Post-Operative Blood Loss
Brief Title: Mechanical Dilatation of the Cervix at Elective Caesarean Section to Reduce Post-Operative Blood Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: cervical dilatation
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Post Operative Hemorrhage
MeSH Terms: conditions — Postoperative Hemorrhage

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: The included patients will be randomized using sealed opaque envelope method into two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (dilation group) (Experimental): the surgeon will perform the cervical dilatation by inserting the double-gloved index ﬁnger into the cervical canal of the patients after the extraction of placenta and membranes. The outer glove will be removed after this procedure. - If failed we will use artery forceps to dilate cervix
  Interventions: Procedure: mechanical dilatation of the cervix
- Group II (non dilatation group) (No Intervention): the surgeon will perform cesarian section without attempting cervical dilatation

INTERVENTIONS:
Procedure: mechanical dilatation of the cervix — the surgeon will perform the cervical dilatation by inserting the double-gloved index ﬁnger into the cervical canal of the patients after the extraction of placenta and membranes. The outer glove will be removed after this procedure.
  - If failed the surgeon will use artery forceps to dilate cervix
  Arms: Group I (dilation group)

SUMMARY:
obstetric hemorrhage remains one of the major causes of maternal death in both developed and developing countries. Because of its importance as a leading cause of maternal mortality and morbidity, and because of evidence of substandard care in the majority of fatal cases, obstetric hemorrhage must be considered as a priority topic for national guideline development.

Some obstetricians believe that the cervix of women at non-labor cesarean section is undilated and might cause obstruction of blood or lochia drainage, leading to postpartum hemorrhage and endometritis from the collection of lochia or debris. Dilatation of the cervix helps with the drainage of blood during postpartum, reducing intrauterine infection or the risk of postpartum hemorrhage. To avoid this problem, some obstetricians routinely dilate the cervix from above during an elective/ non-labor cesarean section using finger, sponge forceps or other instruments

DETAILED DESCRIPTION:
Obstetric hemorrhage remains one of the major causes of maternal death in both developed and developing countries.

Because of its importance as a leading cause of maternal mortality and morbidity, and because of evidence of substandard care in the majority of fatal cases, obstetric hemorrhage must be considered as a priority topic for national guideline development. Obstetric hemorrhage encompasses both antepartum and postpartum bleeding.

The direct pregnancy-related maternal mortality rate in the United States is approximately 7-10 women per 100,000 live births. National statistics suggest that approximately 8% of these deaths are caused by Post Partum Hemorrhage (PPH).

In industrialized countries, PPH usually ranks in the top 3 causes of maternal mortality, along with embolism and hypertension. In the developing world, several countries have maternal mortality rates in excess of 1000 women per 100,000 live births, and World Health Organization statistics suggest that 25% of maternal deaths are due to PPH, accounting for more than 100,000 maternal deaths per year . The most recent Practice Bulletin from the American College of Obstetricians and Gynecologists places the estimate at 140,000 maternal deaths per year or 1 woman every 4 minutes. The rate of PPH increased from 1.5% in 1999 to 4.1% in 2009, and the rate of atonic PPH rose from 1% in 1999 to 3.4% in 2009. In the triennium 2006-2008, 261 women in the UK died directly or indirectly related to pregnancy. The overall maternal mortality rate was 11.39 per 100,000 maternities. Direct deaths decreased from 6.24 per 100,000 maternities in 2003-2005 to 4.67 per 100,000 maternities in 2006-2008 (p = 0.02). The number of deaths from postpartum hemorrhage (PPH) has halved to ﬁve.

In many countries cesarean section (CS) has become the mode of delivery in over a quarter of all births. It is the most commonly performed operation in obstetrics.

Infectious morbidity is the most frequent complication of cesarean delivery. Of women who have caesareans, 5-24% have clinically significant fevers; and 6-21% are diagnosed with uterine infections (endomyometritis or endometritis), 1- 5% with more extensive pelvic infections including abscesses and 2-9% with a breakdown of the surgical incision, most often caused by wound infection. Strategies to minimize postoperative infectious and other morbidities have included modifications of surgical technique, changing of gloves, methods of placental delivery and altering the uterine position during repair of the uterine incision.

However, none of these studies have evaluated the dilatation of the cervix during elective CS. The practice of routine cervical dilatation at elective cesarean section is performed by some surgeons to facilitate discharge of lochia from a uterus that was not in labor in the immediate postoperative period.

A mechanical dilatation of the cervix at cesarean section is deﬁned as an artiﬁcial dilatation of the cervix performed by ﬁnger, sponge forceps or other instruments at non-labor cesarean section.An important concern when dilating the cervix in a non-labor uterus is the theoretical risk of ascending infection to the uterus from the vagina, abdominal cavity and abdominal incision. In addition, cervical dilatation may be associated with the creation of a false passage or hemorrhage from cervical injury. However, an undilated cervix may prevent discharge of lochia following elective CS with retention of lochia, a potential culture medium for bacteria, which can cause puerperal genital tract infection. Some published data from developed countries have suggested that there is no difference in outcome between a practice of routine cervical dilatation or non- dilatation at elective cesarean section.

Turnbull's Obstetrics mentions using an extra glove on the left hand to dilate the cervix. The information currently available about the advantages of cervical dilatation at cesarean section is inconclusive. Therefore, evidence to support the effectiveness or safety of cervical dilatation at cesarean section is needed

.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with a single term fetus >37 weeks of gestational age, with American Society of Anesthesiology (ASA) physical status I or II undergoing Elective Cs (primary or repeated CS).
* Age group 20 - 35 years old

Exclusion Criteria:

* Chorioamnionitis.
* Placenta previa.
* Multiple gestations.
* Preeclampsia.
* Macrosomia.
* Hydramnios.
* Uterine leiomyomata.
* Anemia.
* Previous cervical surgery.
* Previous post-partum hemorrhage.
* Bleeding tendency.
* Hypertension.
* Diabetes mellitus.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 774 (Actual)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Vaginal bleeding during the 1st 24 hours postoperative. | the 1st 24 hours postoperative.
  The amount of vaginal bleeding will be calculated according to number of soaked pads used after the cesarean section for the 1st 24 hours. Where each soaked pad = 50 cc

SECONDARY OUTCOMES:
intraoperative blood loss | during the time of the operation
  Blood loss will be estimated by the anesthesia service to guard against potential surgeon bias.
  Operative blood loss will be calculated from the amount of blood in the suction bottle after delivery of the placenta and the number of towels used and to which degree they were socked.
  Blood from the uterine incision, soaked towels and blood in suction bottle before placental delivery will not be added to the blood measurements.
  Soaked towel = 150 cc. Semi-soaked towel = 75 cc. blood measurements. Soaked towel = 150 cc. Semi-soaked towel = 75 cc.
Total blood loss | operation time plus the 1st 24 hours after operation
  intraoperative blood loss plus potoperative blood loss

CONTACTS AND LOCATIONS:
Overall Officials: mohamed sharkawy, assis.prof., Principal Investigator — Cairo University
Locations (1):
- Faculty of Medicine Cairo University, Cairo, Egypt